CLINICAL TRIAL: NCT02456623
Title: Parent Focused Obesity Intervention for Low-Income African American Preschoolers
Brief Title: Obesity Intervention for Low-Income African American Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Michigan University (Other)
Responsible Party: Principal Investigator, Heather Janisse, Associate Professor, Eastern Michigan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R03DK097444-01 (NIH)
Record Dates: First submitted 2015-01-08; First posted 2015-05-28 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Behavioral intervention that targets the parent of a preschool age child who is overweight. The intervention is 8 sessions in length. Each session is expected to last 1-1.5 hours and will be carried out in the participant's home over 4 months. The sessions will target the nutrition and physical activity knowledge of parents and their motivation for changing parenting related to these factors. Intervention content for the parent will be based on Motivational Interviewing principles.
  Interventions: Behavioral: Intervention
- Attention Control (Active Comparator): The attention control condition includes 1 initial Motivational Interviewing (MI) session conducted in the home. The content of the MI session will be the same as for the intervention participants. Following this session, parents will receive bi-monthly newsletters that will include content similar to what intervention participants receive. AC participants will receive a total of 7 newsletters; 2 on nutrition, 2 on physical activity, 2 on parenting behavior and 1 on community resources. AC participants will also receive a monthly 20-min phone call designed to review newsletter content and answer parent questions.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Intervention — Home-based session targeting the parent
  Arms: Intervention
Behavioral: Attention Control — Attention condition with newsletters and support phone calls
  Arms: Attention Control

SUMMARY:
The purpose of this study is to preliminarily validate a parent-focused obesity intervention program for parents of low-income, African American preschoolers who are currently overweight (> 85th BMI %tile). Half of the participants will receive an intervention that is eight sessions in length and carried out in the participant's home. The sessions will target the nutrition and physical activity knowledge of parents and their motivation for changing parenting related to family eating habits and activity level. The remaining participants will receive an attention comparison control condition (ACCC), which includes one home visit, 7 newsletters and 4 monthly support phone calls. It is hypothesized that children of parents receiving the intervention will have decreases in BMI %tile, consume more fruits/vegetables and fewer sugary beverages, and engage in more activity as compared to ACCC.

DETAILED DESCRIPTION:
This study will do a preliminarily validation of a parent-focused obesity intervention program for parents of low-income, African American preschoolers who are currently overweight (> 85th BMI %tile). Participants will be randomly assigned to an intervention or attention control condition. Those in the intervention will receive an intervention that is eight sessions in length and carried out in the participant's home. The sessions will target the nutrition and physical activity knowledge of parents and their motivation for changing parenting related to family eating habits and activity level. Sessions include psycho-education and skills building exercises. The attention comparison control condition (ACCC) participants will receive one home visit, 7 newsletters and 4 monthly support phone calls. The content of this condition also focuses on nutrition and activity knowledge, motivation and parenting. Outcomes for the intervention and ACC conditions will be assessed at baseline, post-intervention and at a 6-month and 1-year followed up. Child BMI %tile, consumption of fruits/vegetables and sugary beverages, and activity level will be analyzed to examine intervention effectiveness across time.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children enrolled in Head Start preschool in Detroit, MI will be included. Parents must be 18 years of age or older and their child must be of preschool age, between 3 and 5 years of age. Based on recruitment from Detroit Head Start, families will be low-income and of African American descent. Children will have a current body mass index percentile at or above the 85th percentile.

Exclusion Criteria: Child BMI percentile below the 85th percentile.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Child Body Mass Index (BMI) | 5-months
  Change in child BMI will be assessed between baseline and 5-month follow-up.
Change in child fruit, vegetable, and sugary beverage intake using the Block Food Frequency Questionnaire for children | 5-months
  Change in child fruit and vegetable intake between baseline and 5-month follow-up will be collected using the Block Food Frequency Questionnaire for children.
Change in child physical activity level assessed using accelerometers | 5-months
  Change in child's activity level between baseline and 5-month follow-up will be assessed using accelerometers, which will be worn for four days time at each assessment point.

SECONDARY OUTCOMES:
Change in parent nutrition/physical activity knowledge, assessed via a self-report survey | 5-months
  Change in parent knowledge between baseline and 5-month follow-up will be assessed via a self-report survey
Change in parent motivation for health behavior change, assessed using the "readiness ruler" | 5-months
  Change in parent's motivation for health behavior change between baseline and 5-month follow-up will be assessed using the "readiness ruler", which is a self-report survey.
Change in parenting Behavior, assessed using the Caregiver Feeding Style Questionnaire and the Parenting Young Children Scale | 5-months
  Change in parenting behavior between baseline and 5-month follow-up will be assessed using two self-report parent surveys, the Caregiver Feeding Style Questionnaire and the Parenting Young Children Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Heather C Janisse, Ph.D., Principal Investigator — Eastern Michigan University
Locations (1):
- Eastern Michigan University, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No